CLINICAL TRIAL: NCT06607133
Title: Comparison of Staged Thermal Ablation and Thyroidectomy for Large Benign Thyroid Nodules
Brief Title: Thermal Ablation Vs Thyroidectomy for Large Benign Thyroid Nodules
Status: Not yet recruiting | Type: Observational
Sponsor: Ming-an Yu (Other)
Responsible Party: Sponsor-Investigator, Ming-an Yu, Head of the Department of Interventional Medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: S2019-283-02
Record Dates: First submitted 2024-09-08; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-08

CONDITIONS: Benign Thyroid Nodules
Keywords: thermal ablation; Thyroidectomy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- surgery group: patients treated with thyroidectomy for benign thyroid nodules
  Interventions: Procedure: surgery
- thermal ablation group: patients treated with staged thermal ablation for benign thyroid nodules
  Interventions: Procedure: staged thermal ablation

INTERVENTIONS:
Procedure: surgery — patients undergo conventional/open thyroidectomy or endoscopic thyroidectomy for large benign thyroid nodules
  Groups: surgery group
Procedure: staged thermal ablation — patients undergo multiple sessions of thermal ablation for large benign thyroid nodules
  Groups: thermal ablation group

SUMMARY:
To compare the safety, efficacy and quality of life between staged thermal ablation and thyroidectomy in the treatment of Large benign thyroid nodules.

DETAILED DESCRIPTION:
Large benign thyroid nodules （BTNs）usually cause compressive symptoms or cosmetic concerns and therefore require treatment. Thyroidectomy remains the mainstay treatment for large, symptomatic BTNs. However, if surgery is not feasible or refused, ablative approach could be considered in selected patients. However, it has been proved that single application of thermal ablation is less effective in causing shrinkage in large thyroid nodules. The possible reason is that it is difficult for single application of thermal ablation to cover all of the nodule tissue in a three-dimension if the nodule is large. In addition, nodule locations adjacent to vital structures might hinder complete treatment in one session because of safety concerns. Few studies reveal that staged thermal ablation (Pre-designed multiple sessions of thermal ablation) can also achieve complete ablation and adequate volume reduction of large benign thyroid nodules. However, there is a lack of comparison between these two methods. Thus, this study is aimed to compare the safety, efficacy, quality of life between staged thermal ablation and thyroidectomy for treating large benign thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* benign thyroid nodules confirmed by surgical pathology in surgery group, and by two separate US-guided fine-needle aspiration (FNA) or core needle biopsy (CNB) in thermal ablation group;
* the largest diameter of the nodule ≥4 cm;
* the presence of nodule-related symptoms, cosmetic concerns, or psychological stress;
* patients treated with surgery, or staged thermal ablation (who explicitly refused surgery);
* more than 12-month follow-up duration

Exclusion Criteria:

* suspicion of malignant nodule on ultrasound findings (e.g., marked hypoechoic, microcalcifications, or ill-defined margins);
* comorbidities of other severe diseases;
* without complete treatment and/or follow-up information

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated with surgery, or staged thermal ablation in China-Japan Friendship Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
volume reduction ratio | From enrollment to the end of treatment at 12 months
  The volume reduction ratio(VRR) = [(preoperative volume - volume at the follow-up point)/preoperative volume] × 100%. The volumes of the nodules were calculated using the following equation: V=π/6 a×b×c (where V is the volume, a is the maximum diameter, b and c are the other two perpendicular diameters).
Complications | From enrollment to the end of treatment at 12 months
  Complications related to thermal ablation or thyroidectomy during treatment procedures, at the hospital stay and follow-ups.

SECONDARY OUTCOMES:
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire | From enrollment to the end of treatment at 12 months
  Questionnaires of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) was used to evaluate the quality of life for cancer patients. All scales and single-item measures range from score 0-100 after linear transformation. The summary score of QLQ-C30 is used to measure the overall health-related quality-of-life (HRQoL), with a lower score indicating poorer HRQoL. And a higher score on the functional scales and global status scale indicates a better level of functioning and HRQoL, while a higher score on the symptom scales and single item means more discomfort and complaints.
Thyroid Cancer-Specific Quality of Life questionnaire | From enrollment to the end of treatment at 12 months
  The Thyroid Cancer-Specific Quality of Life questionnaire (THYCA-QoL) was used to assess thyroid-specific symptoms in thyroid cancer survivors. The questionnaire consists of seven symptom scales (including neuromuscular, voice, concentration, sympathetic, throat/mouth, psychological and sensory problems) and six single items (including problems with scar, feeling chilly, tingling hands/feet, gained weight, headache, less interest in sex). A higher score on this scale implies more symptoms and complaints.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available because of the patients privacy.